CLINICAL TRIAL: NCT06374030
Title: A Retrospective Study on the Practice and Safety of Airway Management in Dutch Emergency Departments
Brief Title: Retrospective Study of Airway Management in Dutch ED's
Status: Recruiting | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: VieCuri Medical Centre (Other); Catharina Ziekenhuis Eindhoven (Other); Rijnstate Hospital (Other); Zuyderland Medical Centre (Other)
Responsible Party: Principal Investigator, Peter Veldhuis, Principal Investigator, Frisius Medisch Centrum
Other Study IDs: EDSAM2024
Record Dates: First submitted 2024-03-20; First posted 2024-04-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent the intervention of endotracheal intubation: Inclusion criteria:
  All patients who underwent endotracheal intubation between 01-01-2019 and 31-12-2023 in the participating ED's.
  Exclusion criteria:
  Patients for which no information about the intubation can be found in the electronic patient chart will be excluded from the study.
  Interventions: Procedure: Endotracheal intubation

INTERVENTIONS:
Procedure: Endotracheal intubation — All endotracheal intubations carried out in the emergency department of one of the participating hospitals in the time period 01-01-2019 - 31-12-2023

SUMMARY:
Describing characteristics of the practice of airway management in Dutch emergency departments, including information about patient demographics, indications, performer characteristics, equipment and medication used and complications due to intubation.

DETAILED DESCRIPTION:
Endotracheal intubation can be a lifesaving intervention for critically ill patients in the emergency department (ED). Endotracheal intubation is, however, a high-risk procedure with many potential complications, which seem to be even more prevalent when carried out in the ED compared to for example the operating theater. This is possibly due to multiple reasons such as a sicker population, non-elective setting, a higher variability among indications for intubation or competence of providers.

Internationally, large registries were established and multiple observational studies have been performed to gain more information about the methods, safety and complications of intubations in the ED. While in recent years these studies have added to our knowledge of ED airway management, there is still a lack of high-quality studies and there is a strong argument for increased research. To date, no studies have been published of airway management in Dutch EDs. The investigators therefore have no knowledge about any factors possibly influencing intubation outcomes and complications nor comparability with international data. Among these are factors that have been associated with preventable harm and death and insight into these factors could be used for improvement of the safety of airway management in Dutch EDs.

This study is therefore intended to provide a comprehensive review of the clinical practice and characteristics of endotracheal intubations within Dutch EDs. The results could potentially be used for comparative analysis against global datasets. Additionally, the insights gained from this study will shed light on existing gaps prevalent in the current registration processes of intubations in the Netherlands. Furthermore, these insights could act as a stepping stone for future investigations that can lead to a deeper understanding of the methodologies, safety protocols, and associated complications of endotracheal intubations within Dutch EDs

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent endotracheal intubation between 01-01-2019 and 31-12-2023 in the participating ED's

Exclusion Criteria:

* Patients for which no information about the intubation can be found in the electronic patient chart will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent endotracheal intubation between 01-01-2019 and 31-12-2023 in the participating ED's (Leeuwarden Medical Centre, VieCuri Medical Centre, Catharina Hospital, Rijnstate Hospital, Zuyderland Medical Centre)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Different complications of endotracheal intubation | At the time of intervention and consequent 1 hour
  * significant decrease of SpO2. Defined as: desaturation of >10% from baseline or as defined by the treating physician
  * significant decrease of blood pressure. Defined as: systolic pressure <90mmHg with a drop of >20% from baseline or as defined by the treating physician.
  * significant increase of blood pressure. Defined as: systolic pressure > 160mmHg with a rise of >20% from baseline, or as defined by the treating physician.
  * significant bradycardia. Defined as: heart rate < 40/min and a drop of > 20% from baseline, or as defined by the treating physician.
  * significant tachycardia. Defined as: heart rate > 160/min and a rise of > 20% from baseline, or as defined by the treating physician.
  * dental or airway trauma
  * oesophageal or mainstem bronchial intubation
  * vomiting or aspiration
  * laryngospasm
  * equipment failure
  * medication error
  * cardiac arrest
  * failed attempt / need for an emergency surgical airway
  * other

OTHER OUTCOMES:
Intubator characteristics | At the time of intervention and consequent 1 hour
  Specialty and function/seniority of the intubator
Indication for intubation | At the time of intervention and consequent 1 hour
  Indications could be:
  Trauma Burns Drowning Overdose/ingestion Respiratory failure Cardiac arrest (active cardiac arrest) Post-cardiac arrest Stroke Seizure Altered mental status due to other cause (if altered mental status due to stroke, intoxication, seizure or post-cardiac arrest then score as the primary cause) Sepsis Cardiac failure Airway obstruction GI bleed Anaphylaxis Other
Sedation agent used | At the time of intervention and consequent 1 hour
  Ketamine, etomidate, propofol, midazolam
Paralytic agent used | At the time of intervention and consequent 1 hour
  Rocuronium / Succinylcholine
Sedative agent after intubation | At the time of intervention and consequent 1 hour
  Propofol Fentanyl Midazolam Morphine Ketamine Other Not indicated
Method of intubation | At the time of intervention and consequent 1 hour
  Direct laryngoscopy Video (hyperangulated or direct) Fiberoptic Surgical airway
Patient characteristics | At the time of intervention and consequent 1 hour
  Demographics of the patient who underwent endotracheal intubation. Such as age (years), gender (male/female), weight/obesity (BMI)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeuwarden Medical Centre, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT06374030/Prot_SAP_000.pdf